CLINICAL TRIAL: NCT03331939
Title: Effect of Short-term Theta Frequency Stimulation of the Vagus Nerve on Cognition : a Pilot Study
Brief Title: Effect of Short-term Theta Frequency Stimulation of the Vagus Nerve on Cognition in Patients With Refractory Epilepsy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: insufficient study staff
Sponsor: University of California, Davis (Other)
Responsible Party: Principal Investigator, Kiarash Shahlaie, M.D., Ph.D., Associate Professor, University of California, Davis
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 938884
Record Dates: First submitted 2017-11-01; First posted 2017-11-06 (Actual); Last update posted 2017-11-06 (Actual); Status verified 2017-10

CONDITIONS: Refractory Epilepsy
MeSH Terms: conditions — Drug Resistant Epilepsy

STUDY DESIGN:
Intervention Model Description: Pilot Study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- No stimulation (Experimental): All patients will receive three different stimulations
  Interventions: Other: no stimulation
- Beta (25-30 Hz) (Other): Vagal nerve stimulator will be set to Beta (25-30 Hz)
  Interventions: Other: beta (25-30 Hz)
- Theta (5 Hz) (Other): Vagal nerve stimulator will be set to Theta (5 Hz)
  Interventions: Other: Theta (5 Hz)

INTERVENTIONS:
Other: no stimulation — Vagal nerve stimulator will be set to no stimulation
  Arms: No stimulation
Other: beta (25-30 Hz) — Vagal nerve stimulator will be set to beta (25-30 Hz)
  Arms: Beta (25-30 Hz)
Other: Theta (5 Hz) — Vagal nerve stimulator will be set to beta (5 Hz)
  Arms: Theta (5 Hz)

SUMMARY:
The purpose of this investigation is data pilot study of the effect of theta frequency stimulation of the vagus nerve on cognitive performance in patients with refractory epilepsy. We will compare the effects of no stimulation, theta frequency (5 Hz), and 'standard' beta frequency stimulation (25-30 Hz) on cognitive measures. We hypothesize that theta frequency VNS will have a positive effect on memory retention. The goal of this study to provide initial data to inform the design of a larger clinical trial to examine the efficacy of theta VNS.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of Refractory Epilepsy
2. Previously implanted vagal nerve stimulator
3. Willingness and ability to undergo temporary changes to their VNS device settings

Exclusion Criteria:

1. <18 years of age
2. Adults unable to consent
3. Pregnant women
4. Prisoners
5. >20 on the Beck Depression Inventory (BDI)
6. <24 on the Montreal Cognitive Assessment (MOCA)
7. Adults with diagnosis of developmental delay, intellectual disability, or traumatic brain injury (TBI).
8. Adults with reported history of learning disability.
9. Adults unable to use a computer with their dominant hand.
10. Status Epilepticus within the past 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2017-01-06 (Actual); Primary Completion 2017-10-31 (Actual); Study Completion 2017-10-31 (Actual)

PRIMARY OUTCOMES:
California Verbal and Learning Test 2nd edition group 1 | hour 1.5
  Test scored with lower values indicating worse memory and higher values indicating better memory.
  Minimum Value:
  -16
  Maximum Value:
  16
California Verbal and Learning Test 2nd edition group 2 | hour 2.25
  Test scored with lower values indicating worse memory and higher values indicating better memory.
  Minimum Value:
  -16
  Maximum Value:
  16
California Verbal and Learning Test 2nd edition group 3 | hour 3
  Test scored with lower values indicating worse memory and higher values indicating better memory.
  Minimum Value:
  -16
  Maximum Value:
  16

IPD SHARING:
Plan to Share IPD: No